CLINICAL TRIAL: NCT01675492
Title: A Prospective Study to Evaluate the Safety and Effectiveness of Wavefront-Guided LASIK Correction of Mixed Astigmatic Refractive Errors With the iDESIGN Advanced Wavescan Studio™ System and STAR S4 IR™ Excimer Laser System
Brief Title: Safety and Effectiveness of Wavefront-guided LASIK for the Correction of Mixed Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-112-IDMA
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Astigmatism
Keywords: Astigmatism; refractive; error; LASIK
MeSH Terms: conditions — Astigmatism | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- wave-front guided LASIK (Experimental)
  Interventions: Device: LASIK

INTERVENTIONS:
Device: LASIK — Surgeons will perform wavefront-guided LASIK based upon measurements obtained with the iDesign System

SUMMARY:
To demonstrate that wavefront-guided LASIK with measurements from iDesign is safe and effective in the treatment of mixed astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of pre-operative exam
* Best Spectacle Corrected Visual Acuity (BSCVA) of 20/20 or better
* Demonstration of refractive stability
* Anticipated post-operative stromal bed thickness of at lest 250 microns
* Willing and capable of returning for follow-up examinations for the duration of the study

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or intend to become pregnant over the course of the study
* Concurrent use of topical or systemic medications that may impair healing
* History of any medical conditions that could affect wound healing
* History of prior intraocular or corneal surgery, active ophthalmic disease,or other ocular abnormality
* Evidence of keratoconus, corneal irregularity, or abnormal topography in the operative eye(s)
* Known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Hileman, PhD, Study Director — Abbott Medical Optics

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Wave-front Guided LASIK: Vision correction for a mixed astigmatism refraction
Period: Overall Study
Arm/Group | Wave-front Guided LASIK
Started (Number of patients and eyes (units) treated) | 84; 149 eyes
Completed (# subjects and eyes completed 24M visit. 149 eyes of 84 subjects completed 3M visit - approval basis) | 42; 75 eyes
Not Completed | 42; 74 eyes
Not completed — study completed early - product approval | 42

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- Wave-front Guided LASIK: LASIK: Surgeons will perform wavefront-guided LASIK based upon measurements obtained with the iDesign System for mixed astigmatism refraction
Arm/Group | Wave-front Guided LASIK
Number analyzed (Participants) | 84
Number analyzed (eyes) | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 73
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 84

OUTCOME MEASURES:

1. Primary Outcome: Line Loss of More Than Two Lines for Best Spectacle Corrected Visual Acuity (BSCVA)
Description: < 5% of eyes will have a loss of > 2 lines of BSCVA at any postoperative visit, as measured using ETDRS logMAR visual acuity charts at 4 meters
Time Frame: 3 Months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Groups:
- Wave-front Guided LASIK: LASIK: Surgeons will perform wavefront-guided LASIK based upon measurements obtained with the iDesign System for a mixed astigmatism refraction
Arm/Group | Wave-front Guided LASIK
Number analyzed (Participants) | 84
Number analyzed (eyes) | 149
eyes | 149

2. Secondary Outcome: Uncorrected Visual Acuity (UCVA) of 20/40 or Better
Description: 85% of eyes will have UCVA of 20/40 or better, as measured using ETDRS logMAR charts at 4 meters
Time Frame: 3 Months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Wave-front Guided LASIK
Number analyzed (Participants) | 84
Number analyzed (eyes) | 149
eyes | 149

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Wave-front Guided LASIK
All-Cause Mortality (participants affected / at risk) | 0/84
Serious Adverse Events (participants affected / at risk) | 0/84
Other Adverse Events (participants affected / at risk) | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communications prior to public release and can embargo communications regarding trial results at any time.